CLINICAL TRIAL: NCT00378716
Title: A Clinical Trial Comparing Oral Uracil/Ftorafur (UFT) Plus Leucovorin (LV) With 5-Fluorouracil (5-FU) Plus LV in the Treatment of Patients With Stages II And III Carcinoma of the Colon
Brief Title: Combination Chemotherapy in Treating Patients With Resected Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP C-06; U10CA012027 (NIH); NSABP-C-06
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Tegafur; Uracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 5-FU + Leucovorin
  Interventions: Drug: 5-fluorouracil; Drug: leucovorin calcium
- Group 2 (Experimental): Uracil/Ftorarur + leucovorin
  Interventions: Drug: tegafur; Drug: uracil

INTERVENTIONS:
Drug: 5-fluorouracil
  Arms: Group 1
Drug: leucovorin calcium
  Arms: Group 1
Drug: tegafur
  Arms: Group 2
Drug: uracil
  Arms: Group 2

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug is a way to kill more tumor cells.

PURPOSE: Randomized phase III trial to determine the effectiveness of uracil, tegafur,and leucovorin compared with fluorouracil plus leucovorin in patients with resected stage II or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the relative efficacy of oral uracil/tegafur (UFT) with leucovorin (CF) vs. fluorouracil (5-FU) with CF in prolonging overall and disease-free survival in patients with potentially curatively resected stage II/III adenocarcinoma of the colon. II. Compare the prognostic significance of several biomarkers alone or in combination, including DNA mismatch repair gene mutations, p53, deleted colon cancer gene, proliferation status, and thymidylate synthase, in patients treated with UFT/CF vs. 5-FU/CF. III. Evaluate the relationships of various biomarkers to each other and their association with patient and tumor characteristics. IV. Compare quality of life in patients treated with UFT/CF vs. 5-FU/CF.

OUTLINE: This is a randomized study. Patients are stratified by number of positive lymph nodes and participating institution. For the quality-of-life portion of the study, patients are stratified by age, sex, and ethnicity. Treatment begins within 6 weeks after curative resection and within 1 week of randomization. Patients are randomly assigned to one of two groups. The first group receives intravenous leucovorin followed by intravenous fluorouracil weekly for 6 weeks. Treatment repeats every 8 weeks for a total of 3 courses. The second group receives oral uracil/tegafur, and oral leucovorin every 8 hours for 28 days. Treatment repeats every 5 weeks for a total of 5 courses. No concurrent halogenated antiviral agents (e.g., sorivudine) are permitted. After completing treatment, patients complete quality-of-life questionnaires at one year.

PROJECTED ACCRUAL: Approximately 1,500 patients will be entered over 3 years to provide 1,452 evaluable patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the colon that has been curatively resected within 42 days prior to entry, as follows: Stage II (T3-4 N0 M0, Modified Astler-Coller B2/3), i.e., tumor invasion of the wall of the colon or extension into the pericolonic tissue Stage III (any T N1-3 M0), i.e., tumor invasion of any depth No sarcoma, lymphoma, or carcinoid histology No laparoscopically assisted colectomy unless performed on protocol NCCTG-934653 (intergroup study INT-0146) Entire tumor located above the peritoneal reflection on surgical exploration or more than 15 cm from anal verge on endoscopy Involved adjacent structures (e.g., bladder, small intestine, ovary) removed en bloc with histologically negative margins More than 1 synchronous primary colon tumor allowed Most advanced tumor used for stage assignment No previous or synchronous rectal cancer Intestinal obstruction allowed Preliminary or complementary colostomy allowed Walled-off perforation allowed No free perforation, i.e., free air or fluid in abdomen No prior invasive colon or rectal malignancy regardless of disease-free interval

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: At least 10 years (excluding cancer diagnosis) Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST or ALT normal Renal: Creatinine normal Cardiovascular: No active ischemic heart disease No NYHA class III/IV status No myocardial infarction within 6 months No symptomatic arrhythmia within 6 months Other: No nonmalignant systemic disease that precludes protocol treatment No psychiatric or addictive disorder that precludes informed consent No second malignancy within 10 years except: Effectively treated nonmelanomatous skin cancer Surgically cured carcinoma in situ of the cervix Lobular carcinoma in situ of the breast No pregnant women Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1608 (Actual)
Dates: Start 1997-02; Primary Completion 2006-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Compare the relative efficacy of UFT + LV with that of 5-FU + LV in prolonging disease-free survival and survival

SECONDARY OUTCOMES:
evaluate the prognostic significants of proposed biomarkers, alone or in combination, in patients treated with 5-FU + LV or UFT + LV
Evaluate the relationships of various biomarkers to each other and to evaluate their association with patient and tumor characteristics
Compare quality of life in patients with stage II and III carcinoma of the colon treated with either 5-FU + LV or UFT + LV regimen

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. O'Connell, MD, Study Chair — Allegheny Cancer Center at Allegheny General Hospital

REFERENCES:
- [Background] Soran A, Nesbitt L, Mamounas EP, Lembersky B, Bryant J, Anderson S, Brown A, Passarello M. Centralized medical monitoring in phase III clinical trials: the National Surgical Adjuvant Breast and Bowel Project (NSABP) experience. Clin Trials. 2006;3(5):478-85. doi: 10.1177/1740774506070747. PMID 17060221
- [Background] Wang SJ, Zamboni BA, Wieand HS, et al.: Conditional survival for patients with colon cancer: an analysis of National Surgical Adjuvant Breast and Bowel Project (NSABP) trials C-03 through C-06. [Abstract] J Clin Oncol 24 (Suppl 18): A-6005, 302s, 2006.
- [Background] Wolmark N, Colangelo L, Wieand S. National Surgical Adjuvant Breast and Bowel Project trials in colon cancer. Semin Oncol. 2001 Feb;28(1 Suppl 1):9-13. doi: 10.1016/s0093-7754(01)90245-3. PMID 11273592
- [Result] O'Connell MJ, Yothers G, Paik S, et al.: Relationship between tumor gene expression and recurrence in patients with stage II/III colon cancer treated with surgery + 5-FU/LV in NSABP C-06: consistency of results with two other independent studies. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-301, 2008.
- [Result] Kopec JA, Yothers G, Ganz PA, Land SR, Cecchini RS, Wieand HS, Lembersky BC, Wolmark N. Quality of life in operable colon cancer patients receiving oral compared with intravenous chemotherapy: results from National Surgical Adjuvant Breast and Bowel Project Trial C-06. J Clin Oncol. 2007 Feb 1;25(4):424-30. doi: 10.1200/JCO.2005.05.2597. PMID 17264338
- [Result] Lembersky BC, Wieand HS, Petrelli NJ, O'Connell MJ, Colangelo LH, Smith RE, Seay TE, Giguere JK, Marshall ME, Jacobs AD, Colman LK, Soran A, Yothers G, Wolmark N. Oral uracil and tegafur plus leucovorin compared with intravenous fluorouracil and leucovorin in stage II and III carcinoma of the colon: results from National Surgical Adjuvant Breast and Bowel Project Protocol C-06. J Clin Oncol. 2006 May 1;24(13):2059-64. doi: 10.1200/JCO.2005.04.7498. PMID 16648506
- [Result] Soran A, Harlak A, Wilson JW, Nesbitt L, Lembersky BC, Wienad HS, O'Connell MJ. Diverticular disease in patients with colon cancer: subgroup analysis of national surgical adjuvant breast and bowel project protocol C-06. Clin Colorectal Cancer. 2006 Jul;6(2):140-5. doi: 10.3816/ccc.2006.n.031. PMID 16945170
- [Result] Wolmark N, Wieand S, Lembersky B, et al.: A phase III trial comparing oral UFT to FULV in stage II and III carcinoma of the colon: results of NSABP protocol C-06. [Abstract] J Clin Oncol 22 (Suppl 14): A-3508, 247s, 2004.
- [Result] Smith RE, Lembersky BC, Wieand HS, Colangelo L, Mamounas EP. UFT/leucovorin vs 5-FU/leucovorin in colon cancer. Oncology (Williston Park). 2000 Oct;14(10 Suppl 9):24-7. PMID 11098486